CLINICAL TRIAL: NCT04737044
Title: 1: Effects of Antioxidant-rich Sugar as Alternative Compared to Granulated Sugar on Gene Expression and Other Metabolic Parameters in Healthy Subjects 2: Effectiveness of Education Module to Modify Sugar Consumption Among Individuals With Cardio Metabolic Risk
Brief Title: Effects of Antioxidant Sugar vs Granulated Sugar on Metabolic Outcomes in Healthy and Cardio Metabolic Subjects
Acronym: MSS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Termination of study by the Sponsor (Central Sugars Refinery Sdn. Bhd. Malaysia)
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Central Sugars Refinery Sdn Bhd, Malaysia (Unknown)
Responsible Party: Principal Investigator, Barakatun Nisak Bt Mohd Yusof, Associate Professor Dr Barakatun Nisak Mohd Yusof, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MySugarStudy
Record Dates: First submitted 2021-01-15; First posted 2021-02-03 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Gene Expression; Cardiometabolic Risk; Metabolic Syndrome
Keywords: Antioxidant sugar; Gene Expression; Cardio metabolic risks; Education tool
MeSH Terms: conditions — Metabolic Syndrome | interventions — Gene Expression

STUDY DESIGN:
Intervention Model Description: Study 1:
  The study will be using a two-arm single-blinded RCT with 40 subjects in each of the intervention and control groups.
  Study 2:
  The study will be using a three-arm RCT with 23 subjects in each groups (two interventions and one control groups).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Study 1: Normal sugar (No Intervention): Control group will be required to continue consuming normal sugar intake for 8 weeks.
- Study 1:Minimally refined brown sugar (MRBS) (Experimental): Intervention group will be required to consume MRBS as added sugar based on their habitual diet for 8 weeks intervention.
  Interventions: Other: Study 1: MRBS
- Study 2: Normal sugar intake (No Intervention): - The control group will have no intervention and will continue with their normal daily intake for six months.
- Study 2: White sugar (Experimental): * Intervention group I will be advised to reduce sugar intake to no more than 10% from total energy intake.
  * Intervention group I will be given white sugar for daily usage.
  * Participants in this group will be exposed to the nutrition education module (45 minutes per session, once a week) for six months, attend lecture classes and communicate with health educators through communication applications.
  * For the first three months, one-to-one diet counseling will be conducted.
  * Participants' intake of free sugar, as well as other nutrients (carbohydrate, protein, fats, fibre and others) will be closely monitored to ensure compliance to dietary recommendations.
  Interventions: Other: Study 2: White sugar & education module
- Study 2: MRBS (Experimental): * Intervention group II will be advised to reduce sugar intake to no more than 10% from total energy intake.
  * Intervention group II will be given MRBS for daily usage.
  * Participants in this group will be exposed to the nutrition education module (45 minutes per session, once a week) for six months, attend lecture classes and communicate with health educators through communication applications.
  * For the first three months, one-to-one diet counseling will be conducted.
  * Participants' intake of free sugar, as well as other nutrients (carbohydrate, protein, fats, fibre and others) will be closely monitored to ensure compliance to dietary recommendations.
  Interventions: Other: Study 2: MRBS & education module

INTERVENTIONS:
Other: Study 1: MRBS — MRBS as added sugar based on their habitual diet
  Other Names: Food-based and gene expression
  Arms: Study 1:Minimally refined brown sugar (MRBS)
Other: Study 2: White sugar & education module — White sugar for daily usage (<10% daily energy intake)
  Other Names: Food-based and nutrition education study
  Arms: Study 2: White sugar
Other: Study 2: MRBS & education module — MRBS for daily usage (<10% daily energy intake)
  Other Names: Food-based and nutrition education study
  Arms: Study 2: MRBS

SUMMARY:
Study 1: To investigate the effects of antioxidant-rich sugar as alternative compared to granulated sugar on gene expression and other metabolic parameters in healthy subjects.

The hypotheses is antioxidant-rich sugar have positive effects on reducing inflammatory cytokines, oxidative stress biomarkers and other metabolic parameters in intervention group compared to control group.

Study 2: To evaluate the effectiveness of a nutrition education module in modifying sugar consumption and other CMR-related outcomes in individuals with cardiometabolic risk.

The hypotheses is the nutrition education module significantly improves the sugar consumption and other CMR-related outcomes in the intervention groups compared to the control group

DETAILED DESCRIPTION:
Study 1:

After being informed about the study and potential risks, written informed consent will be obtained from all subjects involved in the study. Respondents will be interviewed at Nutritional Status Assessments Lab at University of Putra, Malaysia (UPM) to obtain socio-demographic data, medical status, nutritional status, lifestyle practices and daily dietary intake. This study will be conducted for a period of 8 weeks. The study design is single-blinded parallel-randomized controlled trial (n=80), with 40 subjects in each group (one intervention and one control group). The participants will be selected based on the inclusion and exclusion criteria.

Study 2:

After being informed about the study and potential risks, written informed consent will be obtained from all subjects involved in the study prior to commencing the study. Respondents will be screened at Nutritional Status Assessments Lab at UPM for mental health status, daily sugar intake, cardiometabolic risk factors (waist circumference, blood pressure, fasting blood glucose, triglyceride and high-density lipoprotein cholesterol) where blood pressure and blood sample will be taken by the phlebotomist. Female candidates will be screened for pregnancy or breast feeding. Those who meet the inclusion/exclusion criteria will be selected. They will be informed via communication application whether they are eligible for the study. This study will be conducted for a period of 6 months.

ELIGIBILITY:
Study 1:

Inclusion Criteria:

* Willingness to adhere to study protocol
* Healthy adults to be aged between 18 and 60 years in both genders
* Being non-smoker
* Body mass index (BMI) between 23 - 26.9 kg/m2 (overweight).

Exclusion Criteria:

* Present of any kidney, liver and/or inflammatory disease (inflammatory bowel disease, Rheumatoid arthritis and etc.), thyroid disorder, diabetes (Type 1 & Type 2), cardiovascular or metabolic disease
* Individuals with impaired glucose tolerance or with fasting blood glucose level that more than 5.2 mmol/L
* Pregnancy or lactation
* Alcohol consumption, food allergy
* Individuals who are on regular antioxidant, anti-inflammatory and /or anti-obesity drugs, receiving any glucose lowering and/or lipid lowering medications
* Change in the diet and physical activity (significant weight changes during study period)
* Subjects who habitually consumed beverages rich in sugar such as milo, Teh tarik more than 500 ml, (as tested with the FFQ)

Study 2:

Candidates will be screened for:

* Cardiometabolic risk factors (waist circumference, blood pressure, fasting blood glucose, triglyceride and high-density lipoprotein cholesterol)
* Pregnancy or breast feeding
* Mental health status
* Daily total sugar intake

Inclusion Criteria:

* Malaysian, aged ≥18-59 years old
* Able to read, write and communicate well either in Malay or English
* Attained at least formal education level (secondary school and above)
* Able to use the gadgets and have access to the internet
* Presence with Cardiometabolic risk defines at least any of three out of five risk factors are present and the risk factors are:waist circumference (men: ≥90cm, women:≥80 cm); blood pressure (≥130/85 mmHg); having diabetes mellitus or fasting blood sugar (≥5.6mmol/L); triglyceride (≥1.7 mmol/L) or high-density lipoprotein (men: <1.03 mmol/L, women: <1.3 mmol/L).
* Daily free sugar intake ≥10% of the daily energy intake

Exclusion Criteria:

* Unstable mental health referring to the DASS-21 score for Depression score ≥5; Anxiety score ≥4 and Stress score ≥8 (Ramli, Salmiah, Nurul Ain 2009)
* Uncontrolled type 2 diabetes defines as HbA1c of more than 8% or hypertriglyceridemia of > 10 mmol/L
* Presence with chronic diseases-related complications such as liver disease or stage 3 chronic kidney disease
* Reported abnormal thyroid stimulating hormones
* On current dietary program or medication for weight loss
* On cancer therapy
* Having physical disabilities
* Pregnancy or the desire to become pregnant in the next 3 months

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Study 1: Gene expression of inflammation biomarkers (interleukin-6) | 8 weeks
  Change from baseline in gene expression of interleukin-6 in micrograms at 8th weeks.
Study 1: Gene expression of inflammation biomarkers (TNF-α) | 8 weeks
  Change from baseline in gene expression of TNF-α in picograms per milliliter at 8th weeks.
Study 1: Gene expression of inflammation biomarkers (CPR) | 8 weeks
  Change from baseline in gene expression of CPR in milligram per liter at 8th weeks.
Study 1: Gene expression of oxidative stress biomarkers (MDA) | 8 weeks
  Change from baseline in gene expression of MDA in millimolar at 8th weeks.
Study 1: Gene expression of oxidative stress biomarkers (SOD) | 8 weeks
  Change from baseline in gene expression of SOD in Units per milliliter at 8th weeks.
Study 1: Gene expression of oxidative stress biomarkers (CAT) | 8 weeks
  Change from baseline in gene expression of CAT in nanomoles at 8th weeks.
Study 2: Change from baseline in sugar consumption | 3 months
  Dietary sugar intake will be determined using a 3-day food record and semi-quantitative FFQ of added sugar intake.
  Total sugar (grams per day) in foods will be calculated using formula [(total sugar (grams) - natural sugar (grams)]. The total added sugar intake will be divided into four centiles i.e., 25th percentile [<10.3g (2 tsps.)], 50th percentile [10.3-23.8g (2-5 tsps.)], 75th percentile [23.8-47.0g (5-9 tsps.)] and 100th percentiles [>47g (9 tsps.)].
Study 2: Change from baseline in sugar consumption | 6 months
  Dietary sugar intake will be determined using a 3-day food record and semi-quantitative FFQ of added sugar intake.
  Total sugar (grams per day) in foods will be calculated using formula [(total sugar (grams) - natural sugar (grams)]. The total added sugar intake will be divided into four centiles i.e., 25th percentile [<10.3g (2 tsps.)], 50th percentile [10.3-23.8g (2-5 tsps.)], 75th percentile [23.8-47.0g (5-9 tsps.)] and 100th percentiles [>47g (9 tsps.)].

SECONDARY OUTCOMES:
Study 1: Inflammation biomarkers (interleukin-6) | 8 weeks
  Change from baseline in interleukin-6 in micrograms at 8th weeks.
Study 1: Inflammation biomarkers (TNF-α) | 8 weeks
  Change from baseline in TNF-α in picograms per milliliter at 8th weeks.
Study 1: Inflammation biomarkers (CPR) | 8 weeks
  Change from baseline in CPR in milligram per liter at 8th weeks.
Study 1: Oxidative stress biomarkers (MDA) | 8 weeks
  Change from baseline in MDA in millimolar at 8th weeks.
Study 1: Oxidative stress biomarkers (SOD) | 8 weeks
  Change from baseline in SOD in Units per milliliter at 8th weeks.
Study 1: Oxidative stress biomarkers (CAT) | 8 weeks
  Change from baseline in CAT in nanomoles at 8th weeks.
Study 1: TAC | 8 weeks
  Change from baseline in TAC in millimolar at 8th weeks.
Study 1: Blood pressure | 8 weeks
  Change from baseline in blood pressure in mmHg at 8th weeks.
Study 1: Lipid profile | 8 weeks
  Change from baseline in total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides in mmol/L at 8th weeks.
Study 1: Glucose profile | 8 weeks
  Change from baseline in fasting glucose in mmol/L at 8th weeks.
Study 1: Anthropometric measurements (height) | 8 weeks
  Change from baseline in height in meters at 8th weeks.
Study 1: Anthropometric measurements (weight) | 8 weeks
  Change from baseline in weight in kilograms at 8th weeks.
Study 1: Anthropometric measurements (waist circumference) | 8 weeks
  Change from baseline in waist circumference in centimeters at 8th weeks.
Study 1: Anthropometric measurements (hip circumference) | 8 weeks
  Change from baseline in hip circumference in centimeters at 8th weeks.
Study 1: Body mass index | 8 weeks
  Weight (kg) and height (m) will be combined to report body mass index in kg/m2.
Study 1: Waist hip ratio | 8 weeks
  Waist (cm) and hip circumference (cm) will be combined to report waist hip ratio
Study 1: Change from baseline in sugar consumption at 8th weeks | 8 weeks
  Dietary sugar intake will be determined using a 3-day food record and semi-quantitative FFQ of added sugar intake.
  Total sugar (grams per day) in foods will be calculated using formula [(total sugar (grams) - natural sugar (grams)]. The total added sugar intake will be divided into four centiles i.e., 25th percentile [<10.3g (2 tsps.)], 50th percentile [10.3-23.8g (2-5 tsps.)], 75th percentile [23.8-47.0g (5-9 tsps.)] and 100th percentiles [>47g (9 tsps.)].
Study 1: Change from baseline in physical activity level at 8th weeks | 8 weeks
  - Physical activity level will be measured using International Physical Activity Questionnaire (IPAQ) and results will be categorized as low, moderate and high physical activity.
Study 1: Change from baseline in intensity of physical activity at 8th weeks | 8 weeks
  Metabolic Equivalent Task (minutes/week) will be used to assess the intensity of physical activity.
Study 2: Change from baseline in anthropometric measurements (height) | 3 months
  Height in meters will be taken.
Study 2: Change from baseline in anthropometric measurements (weight) | 3 months
  Weight in meters will be taken.
Study 2: Change from baseline in anthropometric measurements (waist circumference) | 3 months
  Waist circumference in centimeters will be taken.
Study 2: Change from baseline in anthropometric measurements (hip circumference) | 3 months
  Hip circumference in centimeters will be taken.
Study 2: Change from baseline in body mass index | 3 months
  Weight (kg) and height (m) will be combined to report body mass index in kg/m2.
Study 2: Change from baseline in waist hip ratio | 3 months
  Waist (cm) and hip circumference (cm) will be combined to report waist hip ratio.
Study 2: Change from baseline in blood pressure | 3 months
  Blood pressure in mmHg will be taken.
Study 2: Change from baseline in lipid profile | 3 months
  Total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides in mmol/L will be measured.
Study 2: Change from baseline in sugar profile | 3 months
  Fasting glucose in mmol/L will be measured.
Study 2: Change from baseline in antioxidant activity | 3 months
  Antioxidant activity in mmol/L will be measured.
Study 2: Change from baseline in 24-hour urinary sucrose/fructose | 3 months
  Urinary sucrose (mg/day) and fructose (mg/day) will be combined to report 24-hour urinary sucrose/fructose.
Study 2: Change from baseline in knowledge level | 3 months
  Knowledge level of healthy diet and sugar will be tested using Knowledge Assessment Questionnaire. The score will be presented in percentage.
Study 2: Change from baseline in health belief | 3 months
  Health belief model construct will be determined using Health Belief Model questionnaire. Five subscales: perceived susceptibility, perceived severity, perceived benefits, perceived barriers and perceived self-efficacy will be measured and the scores will be presented in percentage.
Study 2: Change from baseline in mental health | 3 months
  Mental health status will be measured using DASS-21 questionnaire, measuring depression (normal cut-off point: 0-4), anxiety (normal cut-off point: 0-3) and stress (normal cut-off point: 0-7).
Study 2: Change from baseline in physical activity level | 3 months
  Physical activity level will be measured using International Physical Activity Questionnaire (IPAQ) and results will be categorized as low, moderate and high physical activity.
Study 2: Change from baseline in intensity of physical activity | 3 months
  Metabolic Equivalent Task (minutes/week) will be used to assess the intensity of physical activity.
Study 2: Change from baseline in anthropometric measurements (weight) | 6 months
  Weight in meters will be taken.
Study 2: Change from baseline in anthropometric measurements (height) | 6 months
  Height in meters will be taken.
Study 2: Change from baseline in anthropometric measurements (waist circumference) | 6 months
  Waist circumference in centimeters will be taken.
Study 2: Change from baseline in anthropometric measurements (hip circumference) | 6 months
  Hip circumference in centimeters will be taken.
Study 2: Change from baseline in body mass index | 6 months
  Weight (kg) and height (m) will be combined to report body mass index in kg/m2.
Study 2: Change from baseline in waist hip ratio | 6 months
  Waist (cm) and hip circumference (cm) will be combined to report waist hip ratio.
Study 2: Change from baseline in blood pressure | 6 months
  Blood pressure in mmHg will be taken.
Study 2: Change from baseline in lipid profile | 6 months
  Total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides in mmol/L will be measured.
Study 2: Change from baseline in sugar profile | 6 months
  Fasting glucose in mmol/L will be measured.
Study 2: Change from baseline in antioxidant activity | 6 months
  Antioxidant activity in mmol/L will be measured.
Study 2: Change from baseline in 24-hour urinary sucrose/fructose | 6 months
  Urinary sucrose (mg/day) and fructose (mg/day) will be combined to report 24-hour urinary sucrose/fructose.
Study 2: Change from baseline in knowledge level | 6 months
  Knowledge level of healthy diet and sugar will be tested using Knowledge Assessment Questionnaire. The score will be presented in percentage.
Study 2: Change from baseline in health belief | 6 months
  Health belief model construct will be determined using Health Belief Model questionnaire. Five subscales: perceived susceptibility, perceived severity, perceived benefits, perceived barriers and perceived self-efficacy will be measured and the scores will be presented in percentage.
Study 2: Change from baseline in mental health | 6 months
  Mental health status will be measured using DASS-21 questionnaire, measuring depression (normal cut-off point: 0-4), anxiety (normal cut-off point: 0-3) and stress (normal cut-off point: 0-7).
Study 2: Change from baseline in physical activity level | 6 months
  Physical activity level will be measured using International Physical Activity Questionnaire (IPAQ) and results will be categorized as low, moderate and high physical activity.
Study 2: Change from baseline in intensity of physical activity | 6 months
  Metabolic Equivalent Task (minutes/week) will be used to assess the intensity of physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiang WL, Mohd Yusof BN, Azlan A, Ismail IZ, Abu Zaid Z. Impacts of a nutrition education intervention in individuals with cardiometabolic risk: Protocol of a randomized controlled trial. Clin Nutr ESPEN. 2022 Jun;49:536-543. doi: 10.1016/j.clnesp.2022.03.037. Epub 2022 Mar 31. PMID 35623864